CLINICAL TRIAL: NCT07242261
Title: Non-invasive Characterisation of Oral Carcinomas in Patients With Fanconi Anaemia
Acronym: Fanc-Oral
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Jean-Godinot (Other)
Collaborators: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025_RIPH_04_Fanc-Oral
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Fanconi Anaemia
Keywords: Fanconi anaemia; oral brushing; head and neck carcinoma
MeSH Terms: conditions — Cystinosis | interventions — Toothbrushing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Fanconi anaemia (Experimental)
  Interventions: Other: Oral brushing

INTERVENTIONS:
Other: Oral brushing — oral brushing of all oral lesions

SUMMARY:
Patients with Fanconi anaemia have an increased risk of developing squamous cell carcinoma of the head and neck. In addition, their genetic vulnerability limits the use of genotoxic treatments such as radiotherapy and chemotherapy, due to increased exposure to severe toxicities.

Less invasive diagnostic techniques, such as brush biopsies, which rely on cytological and ploidy analysis, offer the possibility of more systematic, comprehensive and less painful oral mapping, thereby facilitating earlier diagnosis.

DETAILED DESCRIPTION:
The aim of the study is to investigate the capabilities of oral brushing for the characterisation of oral lesions in patients with Fanconi anaemia.

ELIGIBILITY:
Inclusion Criteria:

* have Fanconi anaemia
* are aged 15 years or older
* have at least one oral lesion with or without warning signs
* who agree to participate in the study

Exclusion Criteria:

* pregnant and breastfeeding women
* protected by law (guardianship, curatorship, judicial protection)
* refusing to participate in the study

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-04-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Oral brushing | Day 0
  * "Positive" result: presence of dysplastic cells at the moderate dysplasia stage or malignant cells.
  * "Negative" result: absence of dysplastic cells beyond the mild dysplasia stage and absence of malignant cells.

SECONDARY OUTCOMES:
oral lesion biopsy | Day 0
  * "Positive" result: presence of dysplastic cells at the moderate dysplasia stage or malignant cells.
  * "Negative" result: absence of dysplastic cells beyond the mild dysplasia stage and absence of malignant cells.